CLINICAL TRIAL: NCT03546738
Title: Spinal Cord Burst Stimulation for Chronic Radicular Pain Following Lumbar Spine Surgery: A Randomized Double-blind Sham-controlled Crossover Trial
Brief Title: Spinal Cord Burst Stimulation for Chronic Radicular Pain Following Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/475
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Back Pain With Radiation; Pain, Postoperative
Keywords: Lumbar Vertebrae; Surgery; Postoperational Complications; Spinal Cord Stimulation
MeSH Terms: conditions — Back Pain; Pain, Postoperative | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the 12 months following implantation of a spinal cord stimulation (SCS) system, the patients will undergo four three-month long periods with either burst SCS or no stimulation (sham) in a randomized order. All patients will undergo two periods of SCS and sham stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Burst SCS (Experimental): Burst Spinal cord stimulation. SCS system implanted and burst stimulation given
  Interventions: Procedure: Burst Spinal Cord Stimulation; Procedure: Sham spinal cord stimulation; Device: SCS implant
- Sham SCS (Sham Comparator): Sham spinal cord stimulation. SCS system implanted but no stimulation given.
  Interventions: Procedure: Burst Spinal Cord Stimulation; Procedure: Sham spinal cord stimulation; Device: SCS implant

INTERVENTIONS:
Procedure: Burst Spinal Cord Stimulation — Burst stimulation utilizes complex programming to deliver high-frequency stimuli of a 40 Hz burst mode with 5 spikes at 500 Hz per spike delivered in a constant current mode
Procedure: Sham spinal cord stimulation — No spinal cord stimulation is provided
Device: SCS implant — a subcutaneously implantable pulse generator ("pacemaker") for long-term therapy.
  The following system from Boston Scientific will be implanted: Precision NoviTM implantable pulse generator and InfinionTM CX 16-contact lead or LinearTM ST 8-contact lead.

SUMMARY:
Spinal cord stimulation (SCS) is a widely applied therapy to treat chronic neuropathic pain, and one of the most common indications is persisting radicular neuropathic pain following lumbar spine surgery. In traditional SCS therapies, the objective has been to replace the pain sensation with paresthesia. The anticipation is that the electrical current alters pain processing by masking the sensation of pain with a comfortable tingling or paresthesia. Although patients mostly cope with paresthesia, a significant proportion reports that the sensation is unpleasant.

'Burst' SCS utilizes complex programming to deliver high-frequency stimuli. This SCS technique seems to provide paresthesia-free stimulation, resulting in better pain relief of low back and leg pain then traditional tonic stimulation.

The widespread use of SCS has not been backed by solid evidence. The absence of placebo-controlled trials has long been an important point of criticism, but due to the nature of the intervention with sensation of paresthesia, studies with placebo control have so far not been considered possible. When 'burst' SCS is used the stimulation is often unnoticed by the patient, allowing comparison with placebo stimulation.

The aim of this randomized double-blind sham-controlled crossover trial is to evaluate the efficacy of 'burst' spinal cord stimulation for chronic radicular pain following spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone ≥1 back surgeries and developed chronic radicular pain that has remained refractory to non-surgical treatment for ≥6 months
* Minimum pain intensity of 5/10 on the leg pain NRS at baseline
* Successful two-week SCS testing period with tonic stimulation (≥2 points reduction in leg pain NRS from baseline). This means patients will experience paresthesia during the SCS trial period
* Mandatory assessment at the Multidisciplinary outpatient clinic for back-, neck- and shoulder rehabilitation, St. Olavs University Hospital

Exclusion Criteria:

* Coexisting conditions that would increase procedural risk (e.g., sepsis, coagulopathy)
* History of laminectomy or posterior fusion at the thoracolumbar junction, where percutaneous electrode end tips are routinely placed.
* Abnormal pain behavior and/or unresolved psychiatric illness.
* Unresolved issues of secondary gain or inappropriate medication use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in disease-specific functional outcome between active burst stimulation and placebo stimulation periods | 12 months
  measured with version 2.0 of the Oswestry disability index (ODI) that has been translated into Norwegian and tested for psychometric properties. The ODI questionnaire quantifies disability for degenerative conditions of the lumbar spine and covers intensity of pain, ability to lift, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. The index is scored from 0 to 100. Zero means no disability and 100 reflects maximum disability.

SECONDARY OUTCOMES:
Change from baseline in generic health-related quality of life measured with the Euro-Qol-5D (5L) between active burst stimulation and placebo stimulation periods | 12 months
Change from baseline in back pain between active burst stimulation and placebo stimulation periods | 12 months
  measured using numerical rating scales (NRS)
Change from baseline in leg pain between active burst stimulation and placebo stimulation periods | 12 months
  measured using numerical rating scales (NRS)
Change from baseline in daily physical activity between active burst stimulation and placebo stimulation periods | 12 months
  measured by use of a body-worn accelerometer (activPALs from PAL Technologies Ltd., Glasgow, United Kingdom) attached by a waterproof tape to the midpoint of the patients' anterior right thigh

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Gulati, md prof, Principal Investigator — St. Olavs Hospital; Geir Bråthen, md prof, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Derived] Hara S, Andresen H, Solheim O, Carlsen SM, Sundstrom T, Lonne G, Lonne VV, Taraldsen K, Tronvik EA, Oie LR, Gulati AM, Sagberg LM, Jakola AS, Solberg TK, Nygaard OP, Salvesen OO, Gulati S. Effect of Spinal Cord Burst Stimulation vs Placebo Stimulation on Disability in Patients With Chronic Radicular Pain After Lumbar Spine Surgery: A Randomized Clinical Trial. JAMA. 2022 Oct 18;328(15):1506-1514. doi: 10.1001/jama.2022.18231. PMID 36255427
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473